CLINICAL TRIAL: NCT06691581
Title: Multicenter Observational Ambispective Study for Congenital Platelet Disorders
Brief Title: Italian Study for Congenital Platelet Disorders
Acronym: SIPaP
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, De Candia Erica, Associate Professor of Internal Medicine, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7003
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: Platelet Disorder
MeSH Terms: conditions — Blood Platelet Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients with established diagnosis will be enrolled.: All patients with established diagnosis of inherited number or function platelet disorder (IPN and IPD, respectively), on the basis of internationally established clinical, laboratory and genetic criteria will be enrolled.

SUMMARY:
Inherited platelet disorders (IPD) are a heterogeneous group of rare bleeding diseases associated with a reduction of platelet number and/or function and with a bleeding tendency ranging from mild to severe. The frequency of inherited thrombocytopenias has been estimated to be 2.7/100,000 while the prevalence of inherited platelet function disorders is unknown, partly because they are frequently overlooked due to their difficult diagnosis.

DETAILED DESCRIPTION:
This a no-profit national multicenter ambispectic (retrospective and prospective) observational study.

After collection of informed consent form each patient, each center will enroll the patient and will collect general, laboratory and clinical data on an electronic CRF on a REDCAP platform. Each patient will receive a unique identification number. All clinical events will be reported in the data base.

ELIGIBILITY:
Inclusion Criteria:

* All patients with established diagnosis of inherited number or function platelet disorder (IPN and IPD, respectively), on the basis of internationally established clinical, laboratory and genetic criteria will be enrolled.
* For patients <18 ys, consensus will be signed by parents or legal responsible

Exclusion Criteria:

* No written consent
* Undocumented or uncertain diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with established diagnosis of inherited number or function platelet disorder (IPN and IPD, respectively), on the basis of internationally established clinical, laboratory and genetic criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
congenital platelet diseases | 48 months
  The main objectives of the study are to collect information on the diagnosis and management of these rare disorders and to create clinical and scientific collaborations between participating centres, and the aim of this project is to create for the first time an ambiseptic multicentre database on clinical and laboratory data on patients with congenital platelet disorders and to observe the prevalence of different congenital platelet disorders

SECONDARY OUTCOMES:
QoL | 48 months
  description of different symptoms and therapeutical options and evaluation of health-related quality of life through validated questionnaires that record the patient's self-assessment of health on a vertical visual analogue scale in which the endpoints are labelled 'best imaginable health' and 'worst imaginable health'

CONTACTS AND LOCATIONS:
Overall Officials: Erica De Candia, MD, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS
Locations (2):
- Italy (2):
  - Fondazione Policlinico Universitario A.Gemelli IRCCS, Roma, Roma
  - Fondazione Policlinico Universitario A.Gemelli IRCCS, Roma, Roma 00168, Rome, rome